CLINICAL TRIAL: NCT07194083
Title: Effectiveness- Implementation Trial of the Function-Based Elopement Treatment
Acronym: (FBET)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mindy Scheithauer, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00009456; 1R34MH136125-01A1 (NIH); 2025P010607 (Other: Emory IRB)
Record Dates: First submitted 2025-09-24; First posted 2025-09-26 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Function Based Elopement Treatment; Autism Spectrum Disorder; Applied Behavior Analysis; Elopement; Functional Analysis
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Cluster Randomization: Random assignment to the treatments, FBET or TAU, will be at the clinic-level, and all participants will receive the intervention to which their respective clinic is assigned.
Who Masked: Outcomes Assessor
Masking Description: Random assignment to the treatments, FBET or TAU, will occur at the clinic level, and all participants will receive the intervention to which their respective clinic is assigned. Randomizations will be blinded to investigators responsible for assessing outcomes (independent evaluators) throughout the study and arranged in a 1:1 ratio (N=3 clinics per intervention, N=6 total) with stratification, ensuring approximately equal representation of clinic sizes (small versus large) between randomized study interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBET: Function-Based Elopement Treatment (Experimental): Clinicals randomized to FBET intervention
  Interventions: Behavioral: Function-Based Elopement Treatment
- TAU: Treatment as Usual (Active Comparator): Clinics randomized to the TAU intervention.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Function-Based Elopement Treatment — FBET is a structured, caregiver-implemented behavioral intervention targeting elopement in children. It includes:
  * Psychoeducation and Behavioral Assessment-caregivers receive training on elopement, behavioral principles, and assessment strategies
  * Functional Analysis Coaching-therapists guide caregivers through a latency-based functional analysis to identify the function of elopement
  * Individualized Treatment Implementation-caregivers apply a function-based plan using differential reinforcement, providing preferred items/activities contingent on safe behavior
  * Treatment Modification-therapists support caregivers in adjusting the plan based on child's response.
  There will be 12 2-hour, caregiver-mediated sessions across 20 weeks Caregivers also learn safety and prevention strategies, including the use of resources like the Big Red Safety Toolkit.
  Other Names: FBET
  Arms: FBET: Function-Based Elopement Treatment
Behavioral: Treatment as Usual — TAU consists of ongoing Applied Behavior Analysis (ABA) services, including caregiver training as it normally exists, provided by the family's Board Certified Behavior Analyst (BCBA), independent of the study protocol. The BCBA determines session frequency, content, and focus based on clinical judgment and the child's individual needs. Topics may include skill acquisition, behavior reduction (including elopement), or other areas deemed relevant to the child's care. The research team does not influence or standardize the TAU content, but will monitor and document the services delivered for descriptive and comparative purposes
  Other Names: TAU
  Arms: TAU: Treatment as Usual

SUMMARY:
The goal of this clinical trial is to test whether the Function-Based Elopement Treatment (FBET) can reduce elopement in children aged 4-12 with autism spectrum disorder (ASD), and to assess its feasibility in community-based Applied Behavior Analysis (ABA) clinics. Researchers will evaluate FBET in a single-arm open-label trial in one clinic, followed by a comparison of FBET to treatment as usual (TAU) across at least six ABA clinics to evaluate effectiveness and implementation.

The main questions it aims to answer are:

* Is it feasible to use FBET in community-based ABA clinics?
* Does FBET reduce elopement?
* Does FBET lead to greater clinical improvement?

Participants will:

* Receive 12 sessions of FBET over 20 weeks with trained BCBAs or receive treatment as usual
* Complete caregiver assessments at baseline and endpoint
* Engage in caregiver training and practice treatment between appointments

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) affects approximately 2.8% of children, or 1 in 36, and is characterized by delayed social communication, restricted interests, and repetitive behaviors. Many children with ASD also exhibit externalizing behaviors such as aggression, self-injury, property destruction, and elopement-defined as leaving supervision without permission. Elopement is a particularly dangerous and stressful behavior, reported as a concern by 35-49% of parents of autistic children. It can occur in various settings, such as bolting in public places or wandering from home, and has been linked to serious injury in nearly 59% of cases. Despite the effectiveness of applied behavior analysis (ABA) strategies in reducing elopement, access to evidence-based treatments (EBTs) remains limited.

The availability of ABA services has grown due to insurance mandates in all 50 states and a significant increase in Board Certified Behavior Analysts (BCBAs), with an estimated 40% of autistic children accessing ABA. However, many BCBAs lack specific training in elopement interventions, such as functional analyses, and only about half provide regular caregiver training. Research has traditionally relied on small-scale studies with limited generalizability and minimal caregiver involvement, creating barriers to widespread implementation.

To address these gaps, researchers developed the Function-Based Elopement Treatment (FBET), a structured, caregiver-mediated ABA intervention designed for real-world settings. FBET includes detailed protocols, decision trees, caregiver scripts, and a workbook to support BCBA implementation and caregiver engagement. In a randomized efficacy trial involving 76 children with ASD and elopement, FBET demonstrated significant improvements over a parent education program (PEP) in reducing elopement severity and frequency, increasing safety measures, and achieving better overall outcomes as rated by independent evaluators.

While FBET shows promise, its effectiveness was tested in a specialized clinic with experienced BCBAs under close supervision. It remains uncertain whether similar results can be replicated in community settings where providers may have less training and support. Nonetheless, FBET represents a meaningful step toward expanding access to effective elopement interventions for children with ASD.

ELIGIBILITY:
Inclusion Criteria:

Child participant:

* Boys and girls ages > 4 to < 12 years
* Autism Spectrum Disorder (ASD) diagnosis by history
* Presence of elopement as an important caregiver concern - elopement occurring regularly for at least 3 months.
* At least one primary caregiver can speak and understand English.

Exclusion Criteria:

• Non-English speaking participants

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in Elopement Questionnaire scores | Baseline, Mid point (8-10 weeks), End point (20 weeks), follow up (32 weeks)
  The Elopement Questionnaire lists situations commonly reported as problematic by caregivers of children with ASD who elope. Aligned with the HSQ, caregivers indicate whether each situation is an issue, and if so, rate the severity from 1 (mild) to 9 (severe). The Elopement Questionnaire creates a total score by summing severity across items.
Feasibility Score Card | Baseline, Mid point (8-10 weeks), End point (20 weeks), follow up (32 weeks)
  This score card includes measures of attendance (BCBAs will keep an attendance log to calculate completed sessions over the expected; score card success = 75% attendance), homework completion (BCBA will score completion ranging from 0 = no to 4 = all homework completed; Success is defined as > 75% of sessions with a score ≥ 3), and therapist integrity (completion of a checklist at a subset of FBET appointments; success defined as >80% accurate implementation) This data will be collected only for the FBET arm

SECONDARY OUTCOMES:
Change in Clinical Global Impression - Improvement (CGI-I) Score | Mid point (8-10 weeks), End point (20 weeks), follow up (32 weeks)
  CGI-I asks an independent evaluator (IE) to rate the degree of improvement, compared to the last visit, on a scale of 1 (very much improved) through 4 (no change) to 7 (very much worse).
Change in Goal Attainment Scaling (GAS) | Baseline, Mid point (8-10 weeks), End point (20 weeks), follow up (32 weeks)
  Goal Attainment Scaling (GAS) will measure appropriate behavior.
  To assess appropriate behavior, at baseline, the independent evaluator (IE) will set 2 goals with the caregiver focused on appropriate behaviors that are relevant for the child's current developmental level. Goals will be weighted by the caregiver. The IE will rate goals at each subsequent assessment visit based on a discussion with the caregiver using a 5-point scale: -2 (worse expected outcome), -1 (less than expected outcome), 0 (expected outcome), +1 (more than expected outcome), and +2 (best expected outcome). Higher the score better the outcome.
Change in Elopement Safety Checklist Score | Baseline, Mid point (8-10 weeks), End point (20 weeks), follow up (32 weeks)
  The Elopement Safety Checklist is a 22-item tool that helps families take steps to prevent elopement and improve safety if it does occur. Items include actions like installing locks or alarms, teaching traffic safety skills, and using identification bracelets. Parents mark "yes" or "no" for each item based on whether it has been completed. The total safety score is calculated as the percentage of items completed-higher scores reflect more safety measures in place to help prevent elopement or protect the child if they elope.

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Scheithauer, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data related to this study will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be entered following standard NDA guidelines, with submissions completed by January 15th and July 15th each year during the study period.
Access Criteria: All of the data is on NDA
URL: https://nda.nih.gov/nda/access-data-info